CLINICAL TRIAL: NCT04987411
Title: Detection of Exhaled Methane Levels for the Recognition and Monitoring of Hemorrhagic Shock - Study Protocol for a Prospective Observational Study
Brief Title: Detection of Exhaled Methane Levels in Hemorrhagic Shock
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, Petra Hartmann MD Ph.D., M.D., Ph.D., Szeged University
Other Study IDs: 5400/2021-SZTE
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Hemorrhagic Shock; Trauma
Keywords: shock; hemorrhagic; methane
MeSH Terms: conditions — Shock, Hemorrhagic; Wounds and Injuries; Shock | interventions — Blood Gas Analysis; Hemodynamic Monitoring; Vital Signs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemorrhagic group: Patients with bleeding confirmed with eFAST or CT.
  Interventions: Diagnostic Test: Measurement of methane concentrations in exhaled breath; Diagnostic Test: Videomicroscopy of the sublingual microcirculation; Diagnostic Test: Blood gas and laboratory analysis; Diagnostic Test: Hemodynamic monitoring

INTERVENTIONS:
Diagnostic Test: Measurement of methane concentrations in exhaled breath — To measure methane concentrations, a near-infrared laser technique-based photoacoustic apparatus will be attached to the exhalation outlet of the ventilator upon arrival of severely injured patients. Exhaled methane levels will be monitored continuously during the first 72 in-hospital hours and will be recorded at pre-determined time points (directly upon arrival, 6 hours post-admission, 12 hours post-admission, 24 hours post-admission, 48 hours post-admission and 72 hours post-admission).
Diagnostic Test: Videomicroscopy of the sublingual microcirculation — Orthogonal polarization spectral imaging technique (Cytoscan A/R, Cytometrics) will be used to visualize the microcirculation of the sublingual mucosa of the patients. The OPS technique utilizes reflected, polarized light at the wavelength of the isobestic point of oxyhemoglobin and deoxyhemoglobin (548 nm). The diminution of sublingual microcirculation can refer to circulatory redistribution due to hemorrhage. Sublingual microcirculation of the patients will be visualized and evaluated at pre-determined time points (directly upon arrival, 6 hours post-admission, 12 hours post-admission, 24 hours post-admission, 48 hours post-admission and 72 hours post-admission) during the first 72 in-hospital hours.
  Other Names: Videomicroscopy using orthogonal polarization spectral imaging (Cytoscan A/R Cytometrics)
Diagnostic Test: Blood gas and laboratory analysis — Arterial blood gas analysis and laboratory testing of venous blood are routine examinations in clinical practice. Base deficit and lactate are considered as global markers of blood loss and shock, and can be obtained rapidly with blood gas analysis. Hemoglobin and hematocrit values can correspond to the severity of blood loss, and are measured routinely both from arterial and venous blood. Sampling of arterial and venous blood for blood gas and laboratory analyses will be performed at pre-determined time points (directly upon arrival, 24 hours post-admission, 48 hours post-admission and 72 hours post-admission) during the first 72 in-hospital hours.
Diagnostic Test: Hemodynamic monitoring — Hemodynamic monitoring is an essential part of emergency trauma care. Non-invasive monitoring of blood pressure, heart rate and respiratory rate of patients will be started immediately upon arrival. After patients are stabilized, invasive arterial blood pressure (IABP) monitoring can be started. IABP is considered as the gold standard of blood pressure measurement in critical care as it reflects the fluctuations of blood pressure in real time. Blood pressure and heart rate values will be recorded at pre-determined time points (directly upon arrival, 6 hours post-admission, 12 hours post-admission, 24 hours post-admission, 48 hours post-admission and 72 hours post-admission) during the first 72 in-hospital hours.
  Other Names: Monitoring vital signs

SUMMARY:
This prospective observational study aims to test the efficacy of the continuous measurement of exhaled methane levels in monitoring the hemodynamic state of severely injured, bleeding trauma patients.

DETAILED DESCRIPTION:
This prospective observational study aims to test the efficacy of the continuous measurement of exhaled methane levels in monitoring the hemodynamic state of severely injured, bleeding trauma patients. Our inclusion criteria require an age of 18 years or greater, an Injury Severity Score (ISS) of 16 or greater, transport directly from scene, intubation on scene or upon arrival, hemorrhage confirmed with eFAST or CT, and signed consent from patient surrogates. Exhaled methane concentrations and indicators of blood loss and shock (vital signs: systolic blood pressure, heart rate; blood gas and laboratory markers: base deficit, lactate, hemoglobin, hematocrit; videomicroscopic image of sublingual microcirculation) will be recorded in pre-determined time points during the first 72 in-hospital hours. The relation between exhaled methane levels and indicators of shock will constitute our primary outcome measures. The association of methane concentrations with clinical outcomes (transfusion need, mortality) will serve as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* injury severity score (ISS)≥16
* intubated on scene or upon arrival
* transported directly from scene to the Emergency Department of the University of Szeged
* hemorrhage confirmed with eFAST or CT
* consent signed by patient surrogate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Severely injured (ISS)≥16, intubated trauma patients with active bleeding.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Association between exhaled methane levels and vital signs | First 72 in-hospital hours
  We intend to investigate the relation between exhaled methane levels and systolic blood pressure and heart rate.
Association between exhaled methane levels and blood gas and laboratory markers | First 72 in-hospital hours
  We intend to investigate the relation between exhaled methane levels and blood gas and laboratory markers (base deficit, lactate, hemoglobin, hematocrit).
Association between exhaled methane levels and sublingual microcirculation | First 72 in-hospital hours
  We intend to investigate the relation between exhaled methane concentrations and sublingual microcirculation.

SECONDARY OUTCOMES:
Association between exhaled methane levels and mortality | First 72 in-hospital hours
  The relation between exhaled methane levels and mortality will be assessed.
Association between exhaled methane levels and number of packed red blood cells required for transfusion/massive transfusion | First 72 in-hospital hours
  The relation between exhaled methane levels and the number of packed red blood cells required for transfusion/massive transfusion will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Traumatology, University of Szeged, Szeged, Hungary

REFERENCES:
- [Background] Barsony A, Vida N, Gajda A, Rutai A, Mohacsi A, Szabo A, Boros M, Varga G, Erces D. Methane Exhalation Can Monitor the Microcirculatory Changes of the Intestinal Mucosa in a Large Animal Model of Hemorrhage and Fluid Resuscitation. Front Med (Lausanne). 2020 Oct 22;7:567260. doi: 10.3389/fmed.2020.567260. eCollection 2020. PMID 33195312
- [Background] Szucs S, Bari G, Ugocsai M, Lashkarivand RA, Lajko N, Mohacsi A, Szabo A, Kaszaki J, Boros M, Erces D, Varga G. Detection of Intestinal Tissue Perfusion by Real-Time Breath Methane Analysis in Rat and Pig Models of Mesenteric Circulatory Distress. Crit Care Med. 2019 May;47(5):e403-e411. doi: 10.1097/CCM.0000000000003659. PMID 30985462
- [Background] Szabo A, Unterkofler K, Mochalski P, Jandacka M, Ruzsanyi V, Szabo G, Mohacsi A, Teschl S, Teschl G, King J. Modeling of breath methane concentration profiles during exercise on an ergometer. J Breath Res. 2016 Feb 1;10(1):017105. doi: 10.1088/1752-7155/10/1/017105. PMID 26828421
- [Derived] Javor P, Rarosi F, Horvath T, Torok L, Varga E, Hartmann P. Detection of exhaled methane levels for monitoring trauma-related haemorrhage following blunt trauma: study protocol for a prospective observational study. BMJ Open. 2022 Jul 6;12(7):e057872. doi: 10.1136/bmjopen-2021-057872. PMID 35793921